CLINICAL TRIAL: NCT03875313
Title: A Phase 1b/2 Open Label, Dose Escalation and Expansion Study of the Glutaminase Inhibitor CB-839 in Combination With the PARP Inhibitor Talazoparib in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study of CB-839 (Telaglenastat) in Combination With Talazoparib in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow Enrollment
Sponsor: Calithera Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CX-839-011
Record Dates: First submitted 2019-03-05; First posted 2019-03-14 (Actual); Results first posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Solid Tumor; Clear Cell Renal Cell Carcinoma; TNBC - Triple-Negative Breast Cancer; Colorectal Cancer; CRC; RCC; ccRCC
Keywords: Tumor Metabolism; Glutaminase Inhibitor; CB-839; telaglenastat; talazoparib; PARP Inhibitor; DNA Damage; DNA Repair; Homologous recombination deficiency; HRD; BRCA 1; BRCA 2
MeSH Terms: conditions — Carcinoma, Renal Cell; Triple Negative Breast Neoplasms; Colorectal Neoplasms | interventions — CB-839; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 600 mg CB-839 + 1 mg Talazoparib (Experimental): 600 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with advanced or metastatic solid tumors.
  Interventions: Drug: CB-839; Drug: Talazoparib
- 800 mg CB-839 + 1 mg Talazoparib: ccRCC (Experimental): 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with incurable/locally advanced or metastatic clear cell renal cell carcinoma (ccRCC) who received ≥ 2 prior systemic regimens including ≥ 1 vascular endothelial growth factor receptor tyrosine kinase inhibitor (VEGFR TKI) therapy.
  Interventions: Drug: CB-839; Drug: Talazoparib
- 800 mg CB-839 + 1 mg Talazoparib: TNBC (Experimental): 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with incurable/locally advanced or metastatic triple-negative breast cancer (TNBC) estrogen receptor (ER)-, progesterone receptor (PR)-, and human epidermal growth factor receptor 2 (HER2)-negative who received ≥ 1 prior line of cytotoxic chemotherapy with no prior poly adenosine diphosphate ribose polymerase (PARP) inhibitor therapy for TNBC or platinum-based chemotherapy for metastatic TNBC.
  Interventions: Drug: CB-839; Drug: Talazoparib
- 800 mg CB-839 + 1 mg Talazoparib: CRC (Experimental): 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with with incurable/locally advanced or metastatic colorectal cancer (CRC) who received appropriate oxaliplatin or irinotecan- and fluorouracil (5-FU)-based chemotherapy with or without bevacizumab.
  Interventions: Drug: CB-839; Drug: Talazoparib
- 800 mg CB-839 + 1 mg Talazoparib: Other Histology (Experimental): 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with other tumor types (prostate, urinary bladder, pancreas, and stomach).
  Interventions: Drug: CB-839; Drug: Talazoparib

INTERVENTIONS:
Drug: CB-839 — CB-839 oral tablets administered twice daily with food at the assigned dose level on 28 day cycles with talazoparib.
  Other Names: telaglenastat
Drug: Talazoparib — Talazoparib oral tablets administered at the standard dose once daily with or without food on 28 day cycles with CB-839.
  Other Names: Talzenna

SUMMARY:
This is a Phase 1b/2 study to determine the recommended phase 2 dose (RP2D), safety and tolerability, pharmacokinetics (PK) and clinical activity of the glutaminase inhibitor CB-839 with the poly adenosine diphosphate ribose polymerase (PARP) inhibitor talazoparib in participants with advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

(Part 1)

-Documented incurable/locally advanced or metastatic solid tumors that have either relapsed or are refractory or intolerant to standard therapies of proven clinical benefit.

(Part 2) Meets 1 of the 3 defined cohorts:

* Cohort 1: Documented incurable/locally advanced or metastatic ccRCC
* Cohort 2: Documented incurable/locally advanced or metastatic defined as ER, PR negative (<1%) and HER2 negative (immunohistochemistry 0 to 1+ or fluorescence in situ hybridization [FISH] negative)
* Cohort 3: incurable/locally advanced or metastatic CRC

For both Parts 1 & 2:

* Recovery to baseline or ≤ Grade 1 Common Terminology Criteria for Adverse Events (CTCAE) v.5.0 from toxicities related to the prior therapy
* Adequate renal, hepatic, and hematological function
* Per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 evaluable disease (Part 1) or measurable disease (Part 2)
* Ability to provide written consent in accordance with federal, local and institutional guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1

Exclusion Criteria for both Parts 1 & 2:

* Prior treatment with CB-839 or a PARP inhibitor
* Unable to received oral medications
* Active and/or untreated central nervous system metastasis. Patients with treated brain metastases must have (1) documented radiographic stability of at least 4 weeks duration demonstrated on baseline central nervous system (CNS) imaging prior to study treatment and (2) be symptomatically stable and off steroids for at least 2 weeks before administration of any study treatment.
* Major surgery within 28 days prior to first dose of study drug
* Receipt of any anticancer therapy within the following windows: small molecule tyrosine kinase inhibitor therapy (including investigational) within the prior 2 weeks or 5 half-lives prior to C1D1, whichever is longer; any type of anti-cancer antibody or cytotoxic chemotherapy within 4 weeks prior to C1D1; radiation therapy for bone metastasis within 2 weeks prior or any other external radiation therapy within 4 weeks prior to C1D1; patients with clinically relevant ongoing complications from prior radiation therapy are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sam Whiting, MD, PhD, Study Director — Calithera Biosciences, Inc
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University, New York, New York
  - MD Anderson, Houston, Texas
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 800 mg CB-839 + 1 mg Talazoparib: TNBC: 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with incurable/locally advanced or metastatic triple-negative breast cancer (TNBC) estrogen receptor (ER)-, progesterone receptor (PR)-, and human epidermal growth factor receptor 2 (HER2)-negativewho received ≥ 1 prior line of cytotoxic chemotherapy with no prior poly adenosine diphosphate ribose polymerase (PARP) inhibitor therapy for TNBC or platinum-based chemotherapy for metastatic TNBC.
Period: Overall Study
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Started | 3 | 16 | 6 | 4 | 4
Completed (All participants discontinued the study, and none entered survival follow up. "Reason Not Completed" presents the reasons for study discontinuation.) | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 16 | 6 | 4 | 4
Not completed — Withdrawal by Subject | 1 | 3 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Study Termination by Sponsor | 0 | 1 | 1 | 0 | 1
Not completed — New Anticancer Treatment | 0 | 1 | 2 | 1 | 0
Not completed — Other, Not Specified | 2 | 11 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- 800 mg CB-839 + 1 mg Talazoparib: ccRCC: 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with incurable/locally advanced or metastatic ccRCC who received ≥ 2 prior systemic regimens including ≥ 1 VEGFR TKI therapy.
- 800 mg CB-839 + 1 mg Talazoparib: TNBC: 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with incurable/locally advanced or metastatic TNBC ER-, PR-, and HER2-negative who received ≥ 1 prior line of cytotoxic chemotherapy with no prior PARP inhibitor therapy for TNBC or platinum-based chemotherapy for metastatic TNBC.
- 800 mg CB-839 + 1 mg Talazoparib: CRC: 800 mg CB-839 taken twice daily and 1 mg talazoparib taken once daily in participants with with incurable/locally advanced or metastatic CRC who received appropriate oxaliplatin or irinotecan- and 5-FU-based chemotherapy with or without bevacizumab.
- Total: Total of all reporting groups
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology | Total
Number analyzed (Participants) | 3 | 16 | 6 | 4 | 4 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (10.00) | 60.8 (10.58) | 51.3 (13.19) | 55.5 (10.66) | 59.0 (11.69) | 58.5 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6 | 2 | 2 | 16
  Male | 3 | 10 | 0 | 2 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 1 | 0 | 3
  Not Hispanic or Latino | 3 | 13 | 6 | 3 | 4 | 29
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 0 | 0 | 2
  Black or African American | 0 | 1 | 2 | 0 | 1 | 4
  White | 2 | 13 | 3 | 4 | 3 | 25
  Other, Not Specified | 0 | 0 | 1 | 0 | 0 | 1
  Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Excluding Deaths Due to Disease Progression
Description: AEs were grades as assessed by CTCAE v 5.0. A TEAE is defined as any AE occurring on or after the first dose of study drug, or existing events that worsened after the first dose during the study, up to 28 days after the last dose.
  An AE is considered "related" if the investigator assessed the relationship as "possibly related" or "probably related." Disease progression includes events in the preferred terms of disease progression and malignant neoplasm progression. Grade 5 disease progression events are excluded from this table.
Time Frame: Start of treatment to 28 days post treatment; mean overall duration of talazoparib exposure was 88.7 days.
Population: Safety Analysis Set: all participants who received at least 1 dose of any study-specific treatment (telaglenastat or talazoparib).
Measure: Count of Participants; unit: Participants
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Number analyzed (Participants) | 3 | 16 | 6 | 4 | 4
Participants
  AE | 3 | 16 | 6 | 3 | 4
  AE grade ≥ 3 | 1 | 12 | 3 | 0 | 3
  AE related to telaglenastat | 3 | 14 | 6 | 2 | 3
  AE related to talazoparib | 3 | 16 | 6 | 2 | 3
  AE related to telaglenastat and talazoparib | 3 | 11 | 6 | 2 | 3
  AE grade ≥ 3 related to telaglenastat | 1 | 4 | 2 | 0 | 1
  AE grade ≥ 3 related to talazoparib | 1 | 11 | 2 | 0 | 2
  AE leading to discontinuation of telaglenastat | 0 | 0 | 0 | 0 | 1
  AE leading to discontinuation of talazoparib | 0 | 0 | 0 | 0 | 1
  AE leading to discontinuation of telaglenastat and talazoparib | 0 | 0 | 0 | 0 | 1
  AE leading to discontinuation of telaglenastat or talazoparib | 0 | 0 | 0 | 0 | 1
  AE leading to telaglenastat dose interruption or reduction | 0 | 10 | 3 | 0 | 4
  AE leading to talazoparib dose interruption or reduction | 1 | 12 | 3 | 0 | 4
  AE leading to telaglenastat and talazoparib dose interruption or reduction | 0 | 9 | 3 | 0 | 4
  AE leading to telaglenastat or talazoparib dose interruption or reduction | 1 | 12 | 3 | 0 | 4
  SAE with CTCAE grade 5 | 0 | 0 | 0 | 0 | 0
  SAE with CTCAE grade 5 related to telaglenastat | 0 | 0 | 0 | 0 | 0
  SAE with CTCAE grade 5 related to talazoparib | 0 | 0 | 0 | 0 | 0
  SAE | 0 | 2 | 1 | 0 | 3
  SAE grade ≥ 3 | 0 | 2 | 1 | 0 | 3
  SAE related to telaglenastat | 0 | 2 | 0 | 0 | 0
  SAE related to talazoparib | 0 | 2 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Laboratory Abnormalities (Hematology, Clinical Chemistry) at More Than 1 Clinic Visit
Description: Hematology parameters conducted included red blood cell (RBC) count, hematocrit, hemoglobin, mean corpuscular volume (MCV), platelet count, white blood cell (WBC) count, neutrophils, lymphocytes, monocytes, eosinophils, and basophils, performed at the discretion of the investigator. Clinical chemistry parameters included aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total bilirubin, direct bilirubin, albumin, total protein, blood urea nitrogen (BUN), creatinine, sodium, potassium, chloride, calcium, carbon dioxide, glucose, and lactate dehydrogenase (LDH), performed at the discretion of the investigator.
Time Frame: Hematology: screening, cycle 1 day 1, cycle 1 day 15, cycle 2 day 1, end of treatment (EOT). Clinical chemistry parameters: screening, cycle 1 day 1, cycle 1 day 8, cycle 1 day 15, cycle 1 day 22, cycle 2 day 1, cycle 2 day 15, EOT.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Number analyzed (Participants) | 3 | 16 | 6 | 4 | 4
Participants
  Hematology | 0 | 0 | 0 | 0 | 0
  Clinical Chemistry | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as an AE determined by the investigator to be possibly or probably related to study drug that also was:
  * Any ≥ Grade (Gr) 4 non-hematological toxicity
  * Gr 3 non-hematologic toxicity, except: fatigue; nausea/vomiting that responds within 24 hours after initiating maximal supportive care; rash or itching that resolves to ≤ Gr 1 within 2 weeks.
  * Any clinically meaningful Gr 3 non-hematologic laboratory value if medical intervention is required OR the abnormality leads to hospitalization, OR the abnormality persists for > 1 week (except Gr 3/4 elevation in serum amylase and/or lipase not associated with clinical or radiological evidence of pancreatitis).
  * Gr ≥ 3 febrile neutropenia
  * Gr ≥ 4 anemia; neutropenia lasting > 7 days; thrombocytopenia
  * Gr 3 thrombocytopenia associated with: a bleeding event that requires a platelet transfusion OR a life-threatening bleeding event occurring due to low platelet count which results in urgent intervention.
Time Frame: During Cycle 1 on Days 1 through 28, inclusive
Population: DLT Evaluable Participants: All participants were considered DLT-evaluable, with the following exceptions: participants who withdrew or were withdrawn from the study prior to completing the DLT assessment window for any reason other than a DLT; participants who did not receive ≥ 75% of the assigned dose (depending on dose level) of telaglenastat and talazoparib, i.e., 42 doses of telaglenastat and 21 doses of talazoparib, in the first 28-day treatment cycle for any reason other than a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Number analyzed (Participants) | 3 | 16 | 6 | 4 | 4
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Overall Response Rate (ORR)
Description: ORR was defined by Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 as the percentage of participants with documented complete response (CR) or partial response (PR) since the date of treatment initiation. CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Stable disease must have been a minimum of 51 days from date of treatment initiation. Exact binomial confidence intervals (Clopper Pearson).
Time Frame: Maximum duration of follow-up for ORR was 12.9 months.
Population: Efficacy Evaluable Population: all participants who had measurable disease at baseline, received at least one dose of study drug (telaglenastat or talazoparib), and completed at least one post-baseline tumor assessment, or discontinued study treatment early due to study drug-related toxicity or for disease-related death.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Number analyzed (Participants) | 2 | 15 | 5 | 4 | 3
percentage of participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]

5. Primary Outcome: Confirmed ORR (cORR)
Description: Overall Response Rate is defined by RECIST v1.1 as the percentage of participants with documented confirmed CR or confirmed PR since the date of treatment initiation. CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR or PR must have been sustained a minimum of 28 days when confirmation was reported. Stable disease must have been a minimum of 51 days from date of treatment initiation. Exact binomial confidence intervals (Clopper Pearson).
Time Frame: Maximum duration of follow-up for cORR was 12.9 months.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Number analyzed (Participants) | 2 | 15 | 5 | 4 | 3
percentage of participants | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 70.8]

6. Primary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate is defined by RECIST v1.1 as the percentage of participants with documented CR, PR, or stable disease (SD) since the date of treatment initiation. CR=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR=At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. CR or PR must have been sustained a minimum of 28 days when confirmation was reported. SD=Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. SD must have been a minimum of 102 days from date of treatment initiation and documented on at least 2 consecutive post-baseline scans. Exact binomial confidence intervals (Clopper Pearson).
Time Frame: Maximum duration of follow-up for CBR was 12.9 months.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Number analyzed (Participants) | 2 | 15 | 5 | 4 | 3
percentage of participants | 0.0 [0.0 to 84.2] | 20.0 [4.3 to 48.1] | 20.0 [0.5 to 71.6] | 0.0 [0.0 to 60.2] | 66.7 [9.4 to 99.2]

7. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from treatment initiation to the date of documented disease progression (PD) within 2 consecutive scheduled radiographic disease assessments or death for any cause, whichever occurs first. PD: ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition, the sum must also demonstrate an absolute increase of ≥ 5 mm. (The appearance of one or more new lesions is also considered progression). Participants with no documentation of PD or death on-study, PD or death occurs after missing 2 consecutive scheduled radiographic disease assessments, or new anti-cancer therapy were censored at the date of last available tumor assessment. Participants missing baseline disease assessments were censored at the date of first dose. Kaplan-Meier product-limit estimates. Brookmeyer-Crowley methodology for a non-parametric 95% CI was used.
Time Frame: Maximum duration of follow-up for PFS was 12.9 months.
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
Number analyzed (Participants) | 2 | 15 | 5 | 4 | 3
months | 1.86 [1.84 to 1.87] | 1.87 [1.77 to 3.88] | 1.71 [1.18 to 3.71] | 1.66 [0.10 to 1.84] | NA [0.92 to NA] — insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: Start of treatment to 28 days post treatment; mean overall duration of talazoparib exposure was 88.7 days.
Description: Per protocol, the serious and nonserious adverse event tables exclude grade 5 disease progression events.
Arm/Group | 600 mg CB-839 + 1 mg Talazoparib | 800 mg CB-839 + 1 mg Talazoparib: ccRCC | 800 mg CB-839 + 1 mg Talazoparib: TNBC | 800 mg CB-839 + 1 mg Talazoparib: CRC | 800 mg CB-839 + 1 mg Talazoparib: Other Histology
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/16 | 0/6 | 0/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/16 | 1/6 | 0/4 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 16/16 | 6/6 | 3/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600 mg CB-839 + 1 mg Talazoparib (N=3) | 800 mg CB-839 + 1 mg Talazoparib: ccRCC (N=16) | 800 mg CB-839 + 1 mg Talazoparib: TNBC (N=6) | 800 mg CB-839 + 1 mg Talazoparib: CRC (N=4) | 800 mg CB-839 + 1 mg Talazoparib: Other Histology (N=4)
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 600 mg CB-839 + 1 mg Talazoparib (N=3) | 800 mg CB-839 + 1 mg Talazoparib: ccRCC (N=16) | 800 mg CB-839 + 1 mg Talazoparib: TNBC (N=6) | 800 mg CB-839 + 1 mg Talazoparib: CRC (N=4) | 800 mg CB-839 + 1 mg Talazoparib: Other Histology (N=4)
Nausea (Gastrointestinal disorders) | 1 | 7 | 4 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 6 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 3 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 11 | 3 | 1 | 2
Pyrexia (General disorders) | 0 | 3 | 0 | 0 | 2
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 10 | 2 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 6 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 4 | 2 | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 4 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 3 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 2 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 5 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypophosphataemia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 3 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Foot fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 1 | 2 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Uterine mass (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication by the PI before either a multi-site publication or 18 months after final multi-site study report. PI can only publish their own results and provide 45 days in advance notice. PI must delete any Calithera confidential information from the publication other than study results and give good faith consideration to other comments made by Calithera. The PI must delay the publication for up to 45 days if requested by Calithera and publicly acknowledge Calithera and Pfizer support.

DOCUMENTS (2):
  • Study Protocol (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03875313/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT03875313/SAP_001.pdf